CLINICAL TRIAL: NCT04266587
Title: Adrenocorticotropic Hormone Stability on Whole Blood
Brief Title: ACTH Stability on Whole Blood
Acronym: STABACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019/0350/HP
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ACTH
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): blood sampling is done on healthy volunteers
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — blood sampling is done on healthy volunteers

SUMMARY:
ACTH is a peptide secreted by pituitary gland and plays an important role in regulating cortisol secretion. ACTH is determined in plasma by immunoassays using specific antibodies. Its determination is difficult because of instability in whole blood. Several factors which influence ACTH stability in blood before analysis have been identified: temperature, hemolysis, time to centrifugation and presence of protease inhibitors. Published results on ACTH whole blood stability seem contradictory.

The objective of this study is to evaluate the effect of aprotinin in 10 healthy volunteers. ACTH measurements will be performed on cobas e602 (Roche Diagnostics, Mannheim, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 to 60,

Exclusion Criteria:

* Adult with insufficient venous capital for blood collection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
ACTH concentration in plasma | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Francois FRAISSINET, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No